CLINICAL TRIAL: NCT03536481
Title: Randomized,Open Label,Two-cycle,Crossover,Single Dose Bioequivalency Study of Two Preparations of Ensartinib Capsules in Healthy Chinese Volunteers Under Fasted State and After Meal
Brief Title: Bioequivalency Study of Ensartinib Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BTP-44315
Record Dates: First submitted 2018-04-15; First posted 2018-05-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T-R cohort under fasted state (Experimental): Subjects will be administered with one single dose of ensartinib capsules (test product) under fasted state, after a wash period of 14 days,the subjects will be administered with one single dose of ensartinib capsules (reference product) under fasted state.
  Interventions: Drug: ensartinib capsules (test product); Drug: ensartinib capsules (reference product)
- R-T cohort under fasted state (Experimental): Subjects will be administered with one single dose of ensartinib capsules (reference product) under fasted state, after a wash period of 14 days,the subjects will be administered with one single dose of ensartinib capsules (test product) under fasted state.
  Interventions: Drug: ensartinib capsules (test product); Drug: ensartinib capsules (reference product)
- T-R cohort after meal (Experimental): Subjects will be administered with one single dose of ensartinib capsules (test product) after meal, after a wash period of 14 days,the subjects will be administered with one single dose of ensartinib capsules (reference product) after meal.
  Interventions: Drug: ensartinib capsules (test product); Drug: ensartinib capsules (reference product)
- R-T cohort after meal (Experimental): Subjects will be administered with one single dose of ensartinib capsules (reference product) after meal, after a wash period of 14 days,the subjects will be administered with one single dose of ensartinib capsules (test product) after meal.
  Interventions: Drug: ensartinib capsules (test product); Drug: ensartinib capsules (reference product)

INTERVENTIONS:
Drug: ensartinib capsules (test product) — Test product(T)：100mg ensartinib capsules manufactured by Betta Pharmaceuticals
  Other Names: X-396 capsules
Drug: ensartinib capsules (reference product) — Reference product(R)：100mg ensartinib capsules manufactured by Catalent Pharma Solutions
  Other Names: X-396 capsules

SUMMARY:
The main objective of this study is to evaluate the bioequivalency of two preparations of ensartinib capsules in Chinese healthy volunteers.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the bioequivalency of two preparations of ensartinib capsules in Chinese healthy volunteers under fasted state or after meal. In addition, the safety of single dose administration of ensartinib capsules in Chinese healthy volunteers will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male body weight≥50.0kg or female body weight≥45.0kg; BMI between 19.0-26.0 kg/m2(inclusive)
* Generally in good health, with no history of chronic disease or sever disease
* No (clinical significant) abnormal findings in clinical laboratory tests and physical examinations
* No plan for pregnancy in coming 6 months, and must practice effective contraception; No plan for sperm or egg donation
* Written informed consent

Exclusion Criteria:

* History of food or drug allergies
* Clinical significant disease or disorders
* Received surgery in 3 months before screening, or have plan for surgery during the study
* Participated in other clinical trials within 3 months before screening
* Venipuncture intolerance
* Drug abusing in 6 months
* Donated ≥200 mL of blood within 30 days before screening
* Pregnant or under lactation period (female subjects)
* Received any prescription drug, over-the-counter drug, Chinese herbal drug or vitamins in 2 weeks
* Received any vaccine in 4 weeks
* Excessively smoking, alcohol or coffin-containing beverage drinking in 3 months
* Other circumstances that is deemed not appropriate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration(Cmax) of ensartinib(test product) after meal | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The Cmax of ensartinib(test product) in after meal blood samples of each subject over a 120 hour period post dose
Peak plasma concentration(Cmax) of ensartinib(test product) under fasted sate | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The Cmax of ensartinib(test product) in fasting blood samples of each subject over a 120 hour period post dose
Peak plasma concentration(Cmax) of ensartinib(reference product) after meal | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The Cmax of ensartinib(reference product) in after meal blood samples of each subject over a 120 hour period post dose
Peak plasma concentration(Cmax) of ensartinib(reference product) under fasted sate | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The Cmax of ensartinib(reference product) in fasting blood samples of each subject over a 120 hour period post dose
Area under the plasma concentration versus time curve(AUC) of ensartinib(test product) after meal | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The AUC of ensartinib(test product) in after meal blood samples of each subject over a 120 hour period post dose
Area under the plasma concentration versus time curve(AUC) of ensartinib(test product) under fasted sate | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The AUC of ensartinib(test product) in fasting blood samples of each subject over a 120 hour period post dose
Area under the plasma concentration versus time curve(AUC) of ensartinib(reference product) after meal | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The AUC of ensartinib(reference product) in after meal blood samples of each subject over a 120 hour period post dose
Area under the plasma concentration versus time curve(AUC) of ensartinib(reference product) under fasted sate | pre-dose(60minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The AUC of ensartinib(reference product) in fasting blood samples of each subject over a 120 hour period post dose

SECONDARY OUTCOMES:
Percentage of participants with adverse events as assessed by CTCAE v4.03 | from screening to post-study visit, assessed up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Zhu, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China